CLINICAL TRIAL: NCT03123159
Title: Clinical Utility of the DxN HBV Assay as an Aid in the Management of HBV-Infected Individuals Undergoing Antiviral Therapy
Brief Title: Clinical Performance Evaluation of DxN HBV Assay
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HBV-02-13
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen plasma samples are retained for this study and possible future studies.
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- HBV Infected patients: chronic HBV patients who will undergo standard of care FDA approved antiviral therapy to treat HBV infections. Will have blood drawn to be tested using the DxN HBV Assay. Study is observational and results will not be used to manage patient care.
  Interventions: Diagnostic Test: DxN HBV Assay

INTERVENTIONS:
Diagnostic Test: DxN HBV Assay — Molecular diagnostic test to detect Hepatitis B

SUMMARY:
The DxN Hepatitis B Virus (HBV) Assay is an in vitro diagnostic assay intended as an aid in the management of HBV-infected individuals undergoing antiviral therapy. The purpose of the study is to establish the clinical performance of the DxN HBV Assay for plasma samples in the intended use population.

DETAILED DESCRIPTION:
Same as brief summary.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has serological evidence of chronic HBV infection, and measurable HBV-DNA and ALT at baseline
* Subject will undergo treatment with tenofovir or entecavir for a minimum of 48 weeks

Exclusion Criteria:

* Co-infection with HIV or HCV at enrollment
* Subject has decompensated liver disease or liver cancer
* Prior participation in study
* Current or planned participation in an investigational drug or device study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older with chronic HBV who will undergo antiviral therapy to treat HBV infections
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | Up to 48 weeks
  Defined as unquantifiable HBV Viral load at 48 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lofaro, MSHS, Study Chair — Beckman Coulter
Locations (10):
- United States (8):
  - Scripps Clinic, La Jolla, California
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - Albert Einstein Medical School, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington / Harborview Medical Center, Seattle, Washington
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Centre Hospitalier de l'universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No